CLINICAL TRIAL: NCT02963038
Title: Autologous CD19-targeting CAR T Cells for Refractory B Cell Malignancy
Brief Title: CAR T Cells for Refractory B Cell Malignancy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SenL_19
Record Dates: First submitted 2016-10-28; First posted 2016-11-15 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2016-11

CONDITIONS: B-Cell Leukemia; B-Cell Lymphoma
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CD19 CAR T cells (Experimental): Autologous CD19-targeting CAR T cells
  Interventions: Biological: Autologous CD19-targeting CAR T cells

INTERVENTIONS:
Biological: Autologous CD19-targeting CAR T cells — Autologous CD19-targeting CAR T cells with three signaling domains derived from CD3zeta, CD28 and 4-1BB.

SUMMARY:
Chimeric antigen receptor (CAR) T cells targeting CD19 will be evaluated for safety and efficacy in patients with B cell malignancy including lymphoma or leukemia.

DETAILED DESCRIPTION:
The CAR consists of a CD19 targeting antibody scFv with three intracellular signaling domains derived from CD3 zeta, CD28 and 4-1BB. Autologous T cells will be gene engineered with the CAR gene using a lentivirus vector. Prior to T cell infusion, the patients will be subjected to preconditioning treatment. After T cell infusion, the patients will be evaluated for 24 months for adverse reactions, persistence of CAR T cells and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. The treat history meeting the following criteria:

   * Recurrence of lymphoma patients with imaging (CT/MRI/PET-CT) detection and pathological diagnosis, or recurrence including bone marrow morphology relapse and the MRD recurrence of myeloma patients or leukemia patients, after chemotherapy or stem cell transplantation;
   * Can't get complete remission (including MRD positive) after more than twice repeated chemotherapy of incipient lymphoma, myeloma or leukemia patients;
   * One or twice chemotherapy cannot get remission again (including MRD positive), but not suitable for chemotherapy of incipient lymphoma, myeloma or leukemia patients.
2. There is a measurable lesions before treatment at least;
3. ECOG score≤2;
4. To be aged 1 to 70 years;
5. More than a month lifetime from the consent signing date

Exclusion Criteria:

* Serious cardiac insufficiency, left ventricular ejection fraction<50;
* Has a history of severe pulmonary function damaging;
* Merging other malignant tumor;
* Merging uncontrolled infection;
* Merging the metabolic diseases (except diabetes);
* Merging severe autoimmune diseases or immunodeficiency disease;
* patients with active hepatitis B or hepatitis C;
* patients with HIV infection;
* Has a history of serious allergies on Biological products (including antibiotics);
* Happened in 3 ~ 4 acute GvHD after allogeneic hematopoietic stem cell transplantation on recurring patients Pregnancy or lactation women; Any situation that would increase dangerousness of subjects or disturb the outcome of the clinical study according to the researcher's evaluation.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Tumor load | Up to 24 months
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis.

SECONDARY OUTCOMES:
CAR T cell persistence | Up to 24 months
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis

OTHER OUTCOMES:
B cell number and immunoglobulins in peripheral blood | Up to 12 months
  The number of B cells and immunoglobulins in peripheral blood will be evaluated by routine methods

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Luo, PhD & MD, Principal Investigator — The Second Hospital of Hebei Medical University
Locations (1):
- No.2 Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No